CLINICAL TRIAL: NCT01639443
Title: Reducing VA No-Shows: Evaluation of Predictive Overbooking Applied to Colonoscopy
Acronym: No-show
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 12-055; 1I01HX000878-01 (NIH)
Record Dates: First submitted 2012-07-09; First posted 2012-07-12 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Colon Cancer
Keywords: quality improvement; Organization and Administration; Costs and cost analysis; Patient satisfaction; Health plan implementation
MeSH Terms: conditions — Colonic Neoplasms; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fast-tracked (Experimental): 'Predictive no-show overbooking' intervention. Patients who volunteer to enroll in "fast-track" line, which gives them an opportunity to overbook their appointment for endoscopy earlier in a predictive no-show slots.
  Interventions: Other: Predictive no-show overbooking
- Control (No Intervention): Patients who are scheduled routinely

INTERVENTIONS:
Other: Predictive no-show overbooking — During intervention period, every Veteran scheduled for an endoscopy will be offered "fast-track" offer, which gives them a chance to get their endoscopy procedure done earlier than usual scheduling by overbooking their appointment in a predictive no-show slot.
  Arms: Fast-tracked

SUMMARY:
In this research study, investigators use colonoscopy as a case example to evaluate a predictive overbooking model derived using patient-level predictors of absenteeism. The no-show overbooking intervention employs a logistic regression model that uses patient data to predict the odds of no-showing with 80% accuracy. These projected no-show appointments will be overbooked by clerks for patients who agree to join a "fast track" short-call line. By rapidly processing endoscopy patients and moving them out of traditional slots, investigators predict more scheduling slots would become available for patients awaiting colonoscopy.

DETAILED DESCRIPTION:
Patient "no-shows" are especially common in VA gastrointestinal (GI) endoscopy units, where both open-access endoscopy scheduling and patient dislike of procedures contribute to high absenteeism. In this proposal, investigators use endoscopy as a case example to evaluate a predictive overbooking model derived using patient-level predictors of absenteeism. The no-show overbooking intervention employs a logistic regression model that uses patient data to predict the odds of no-showing with 80% accuracy. These projected no-show appointments will be overbooked by clerks for patients who agree to join a "fast track" short-call line. However, patients scheduled for upper endoscopies in the "fast track" assume a small risk of service denial on the day of their overbooking in case of inaccurate predictions. If this occurs, the patient is guaranteed service in the next available position and is assured of having a shorter wait time. Patients scheduled for colonoscopies will never be turned down but may experience delays in the waiting room the day of their "fast track" appointment. By rapidly processing endoscopy patients and moving them out of traditional slots, investigators predict more scheduling slots would become available for patients awaiting colonoscopy. Investigators propose to conduct a prospective, 24-month, interrupted time series (ITS) trial in the WLAVA (West Los Angeles Veterans Administration) GI clinic endoscopy unit. During intervention periods, investigators will activate the no-show predictive overbooking strategy described above. Investigators will compare outcomes between scheduling strategies, including differences in percent utilization of capacity (primary outcome), number of Veterans served, mean patient lag time between scheduling and procedure, number of unexpected service denials ("bumps") from no-show predictive overbooking, and direct costs of care. Investigators will analyze differences using both traditional univariate and multivariate approaches, and using autoregressive integrated moving average (ARIMA) analyses to adjust for auto-correlations in ITS data.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for upper endoscopy and agree to the terms of "fast track" offer.

Exclusion Criteria:

* If a patient expresses concern about service denial, confusion about the bargain, or refuses to participate, the investigators will schedule these patients routinely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-07-08 (Actual); Primary Completion 2015-07-06 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul G. Shekelle, MD PhD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reid MW, Cohen S, Wang H, Kaung A, Patel A, Tashjian V, Williams DL Jr, Martinez B, Spiegel BM. Preventing patient absenteeism: validation of a predictive overbooking model. Am J Manag Care. 2015 Dec;21(12):902-10. PMID 26671702
- [Result] Reid MW, May FP, Martinez B, Cohen S, Wang H, Williams DL Jr, Spiegel BM. Preventing Endoscopy Clinic No-Shows: Prospective Validation of a Predictive Overbooking Model. Am J Gastroenterol. 2016 Sep;111(9):1267-73. doi: 10.1038/ajg.2016.269. Epub 2016 Jul 5. PMID 27377518
- [Result] May FP, Reid MW, Cohen S, Dailey F, Spiegel BM. Predictive overbooking and active recruitment increases uptake of endoscopy appointments among African American patients. Gastrointest Endosc. 2017 Apr;85(4):700-705. doi: 10.1016/j.gie.2016.09.001. Epub 2016 Sep 10. PMID 27623103

RESULTS

PARTICIPANT FLOW:
Groups:
- Fast-tracked: Patients who volunteer to enroll in "fast-track" line, which gives them an opportunity to overbook their appointment for endoscopy earlier in a predictive no-show slots.
  Predictive no-show overbooking: During intervention period, every Veteran scheduled for an upper endoscopy will be offered "fast-track" offer, which gives them a chance to get their endoscopy procedure done earlier than usual scheduling by overbooking their appointment in a predictive no-show slot.
Period: Overall Study
Arm/Group | Fast-tracked | Control
Started | 180 (These individuals opted into Fast-tracked group and were consented.) | 4855 (These individuals opted to not participate in Fast-tracked group, and were not consented.)
Completed | 180 (Intervention is limited to appointment booking, and all completed.) | 4855 (These individuals all booked appointments using typical booking.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Participants in all study phases.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fast-tracked | Control | Total
Number analyzed (Participants) | 180 | 4855 | 5035
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 112 | 2812 | 2924
  >=65 years | 68 | 2043 | 2111
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (13.6) | 62.2 (10.0) | 62.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 206 | 218
  Male | 168 | 4649 | 4817
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 565 | 582
  Not Hispanic or Latino | 163 | 4290 | 4453
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 35 | 37
  Asian | 5 | 109 | 114
  Native Hawaiian or Other Pacific Islander | 2 | 28 | 30
  Black or African American | 70 | 1584 | 1654
  White | 83 | 2414 | 2497
  More than one race | 2 | 41 | 43
  Unknown or Not Reported | 16 | 644 | 660
Region of Enrollment [Number; unit: participants]
  United States | 180 | 4855 | 5035

OUTCOME MEASURES:

1. Primary Outcome: Percentage of GI Clinic Capacity Filled
Description: Investigators' primary objective will be to evaluate the impact of no-show predictive overbooking on percentage of the GI endoscopy clinic that are filled on a given day. Days where at least one Fast-tracked patient attended an appointment were compared to days where only Control patients attended appointments. Percentage of GI Clinic Capacity is calculated as the number of appointments completed divided by number of appointment spots available on a given day. This percentage was compared between Fast-tracked days and Control days, using data from 1672 patients.
Time Frame: After 12 months of running study in clinic
Population: These 1672 patients are a subset of all patients who were enrolled in this study. We dropped data on a first wave of participants (69 Fast-tracked and 3294 Controls) because of problems incorporating recruitment strategy into clinic. However, data from these individuals was used to build predictive model.
Measure: Mean (Standard Deviation); unit: percentage of clinic capacity filled
Arm/Group | Fast-tracked | Control
Number analyzed (Participants) | 111 | 1561
percentage of clinic capacity filled | 99.6 (19.4) | 86.4 (21.6)
Statistical Analysis 1: Comparison: Fast-tracked vs Control; We counted days containing at least one Fast-tracked participant as a "Fast-tracked" day for the sake of analysis at the clinic level. Our null hypothesis is that these days will not differ in terms of percentage of clinic capacity filled. We are powered to detect a 0.5 Standard Deviation (SD) difference in clinic capacity (Type I error rate = 5%; Power = 81%), with a equal ratio of Experimental and Control days; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Scheduling-to-procedure Lag Time
Description: The investigators will calculate the mean daily lag time for all colonoscopy and upper endoscopies performed per day
Time Frame: After 12 months of running study in clinic
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fast-tracked | Control
Number analyzed (Participants) | 111 | 1561
days | 8.3 (24.3) | 10.8 (24.0)
Statistical Analysis 1: Comparison: Fast-tracked vs Control; We calculated this measure on the patient level. Our null hypothesis is that the lag time between scheduling and appointment, measured in days, will not differ between groups. We are powered to detect a 0.3 SD difference in lag time (Type I error rate = 5%; Power = 84%), accounting for the large sampling ratio (approximately 14:1); Test type: Superiority or Other; p = 0.29, t-test, 2 sided

3. Secondary Outcome: Daily Service Denials ("Bumps")
Description: The investigators will compare the number of patients bumped per day between scheduling approaches
Time Frame: After 12 months of running study in clinic
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fast-tracked | Control
Number analyzed (Participants) | 111 | 1561
participants | 0 | 29
Statistical Analysis 1: Comparison: Fast-tracked vs Control; We did not explicitly power this study to detect differences in the number of service bumps, but we can compare them using Fisher's Exact Test; Test type: Superiority or Other; p = 0.49, Fisher Exact — We would have only expected 2 patients to be bumped in the Experimental Group, and observed 0

4. Secondary Outcome: Advanced Adenoma Detection/Cecal Intubation Rates
Description: The investigators will compare daily advanced adenomatous polyp detection and daily cecal intubation rates between groups.
Time Frame: After 20 months of running study in clinic
Population: We only collected data on polyp detection for the first half of our Fast-tracked participants and all Controls seen over the same time period (4897 in total).
Measure: Mean (Standard Deviation); unit: Number of Polyps Detected per patient
Arm/Group | Fast-tracked | Control
Number analyzed (Participants) | 90 | 4807
Number of Polyps Detected per patient | 2.35 (1.58) | 2.88 (2.56)
Statistical Analysis 1: Comparison: Fast-tracked vs Control; We calculated this measure on the patient level, but were hampered by a large sampling ratio (more than 50:1). Our null hypothesis is that the number of polyps detected will not differ between groups. We are powered to detect a 0.25 SD difference in polyp count per patient (Type I error rate = 5%; Power = 80%); Test type: Superiority or Other; p = 0.05, t-test, 2 sided

5. Secondary Outcome: Length of Workday
Description: Length of Workday in hours (comparing days with Fast-Tracked Appointments to Control days without)
Time Frame: After 12 months of running study in clinic
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fast-tracked | Control
Number analyzed (Participants) | 111 | 1561
hours | 8.31 (1.32) | 7.84 (1.32)
Statistical Analysis 1: Comparison: Fast-tracked vs Control; We counted days containing at least one Fast-tracked participant as a "Fast-tracked" day for the sake of analysis at the clinic level. Our null hypothesis is that these days will not differ in terms of length of workday. We are powered to detect approximately 0.5 SD difference in workday length in hours (Type I error rate = 5%; Power = 81%), with a equal ratio of Experimental and Control days; Test type: Superiority or Other; p = 0.024, t-test, 2 sided

6. Secondary Outcome: Cost Comparisons
Description: For cost comparisons, the investigators will aggregate total provider overtime costs for colonoscopies performed. Cost is reported per day.
Time Frame: After 12 months of running study in clinic
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Fast-tracked | Control
Number analyzed (Participants) | 111 | 1561
dollars | 63.01 (107.01) | 36.88 (101.73)
Statistical Analysis 1: Comparison: Fast-tracked vs Control; We counted days containing at least one Fast-tracked participant as a "Fast-tracked" day for the sake of analysis at the clinic level. Our null hypothesis is that these days will not differ in terms of cost per day. We are powered to detect a 0.5 SD difference in clinic capacity (Type I error rate = 5%; Power = 81%), with a equal ratio of Experimental and Control days; Test type: Superiority or Other; p = 0.11, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: After 24 months of running study in clinic
Description: This study involved scheduling patients for appointments, so the odds of an adverse event are extremely low.
Arm/Group | Fast-tracked | Control
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/4855
Other Adverse Events (participants affected / at risk) | 0/180 | 0/4855

LIMITATIONS AND CAVEATS:
This study was impeded by our ability to schedule Veterans into Fast-Tracked appointments. Although the method is very promising, integration of predictive scheduling is vital for this program to benefit Veterans on a large scale.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes